CLINICAL TRIAL: NCT04191057
Title: Normal Range Study for Free Light Chains in Blood Among Identical or Fraternal Twins
Brief Title: Determining Normal Range for Free Light Chains in Serum Among Twins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-25508
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: free light chains; healthy twins
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Masking Description: The participant will not be given the results of the free light chain result
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy twin (Experimental): Free light chains of twins compared to non-twin siblings
  Interventions: Other: Free light chains

INTERVENTIONS:
Other: Free light chains — Blood samples will be collected and analyzed

SUMMARY:
The objective of this study is to recruit healthy adult identical and fraternal twins for the collection of one teaspoon of blood to be sent to the Clinical Lab at San Francisco General Hospital. The serum will be tested to determine the reference range for free light chains.

DETAILED DESCRIPTION:
Serum free light chains are used to assist in the diagnosis of multiple myeloma. The test measures kappa (K) and lambda (L) chains, and the calculation of the ratio of kappa to lambda (K/L). Previous studies have shown that the K/L ratio does not change over time (1 year). The hypothesis of this study is that healthy twins will have a K/L ratio that are close to each other in value, suggesting that this ratio is genetically linked.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects 18-80 years.
* Must be an identical or fraternal twin (both must be recruited)

Exclusion Criteria:

* Symptoms suggestive of multiple myeloma (e.g., renal insufficiency, anemia, bone pain) -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Free light chain reference range | One month after the completion of the enrollment
  Determination of the normal range for free light chains

CONTACTS AND LOCATIONS:
Overall Officials: Alan Wu, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Participants and other researchers will not have access to data.

REFERENCES:
- [Background] Braga F, Infusino I, Dolci A, Panteghini M. Biological variation of free light chains in serum. Clin Chim Acta. 2013 Jan 16;415:10-1. doi: 10.1016/j.cca.2012.09.008. Epub 2012 Sep 11. No abstract available. PMID 22981867
- [Background] Katzmann JA, Clark RJ, Abraham RS, Bryant S, Lymp JF, Bradwell AR, Kyle RA. Serum reference intervals and diagnostic ranges for free kappa and free lambda immunoglobulin light chains: relative sensitivity for detection of monoclonal light chains. Clin Chem. 2002 Sep;48(9):1437-44. PMID 12194920